CLINICAL TRIAL: NCT05934864
Title: Different Molecular Subtypes of Peripheral T-cell Lymphoma, a Real-world Registry Study. (TRUST Study)
Brief Title: Different Molecular Subtypes of Peripheral T-cell Lymphoma, a Real-world Registry Study. (TRUST)
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: West China Hospital (Other); Shandong Provincial Hospital (Other Government); RenJi Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Deputy Director of Hospital, Shanghai Rui Jin Hospital, Ruijin Hospital
Other Study IDs: RJ-PTCL-3
Record Dates: First submitted 2023-06-13; First posted 2023-07-07 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Peripheral T Cell Lymphoma; molecular subtypes
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Targeted sequencing was performed in fresh tissue or FFPE tissue quality controlled.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gene mutation profile of PTCL: 84-gene penal was targeted sequenced in 1000 PTCL patients to investigate their mutation profile and molecular subtypes.
  Interventions: Genetic: 84-gene penal

INTERVENTIONS:
Genetic: 84-gene penal — 84-gene penal was targeted sequenced in 1000 PTCL patients to investigate their mutation profile and molecular subtypes.

SUMMARY:
A multi-center, prospective, registry study to analyze the clinical characteristics and prognosis of different molecular subtypes of peripheral T-cell lymphoma.

DETAILED DESCRIPTION:
Peripheral T-cell lymphoma (PTCL）is a distinct and heterogeneous histopathologic subtype of non-Hodgkin lymphoma (NHL), accounting for ~10%. Patients with PTCL still have poor treatment response and prognosis under conventional CHOP regimen. This multi-center, prospective, registry study is designed to analyze the clinical characteristics and prognosis of different molecular subtypes of PTCL. The results can guide future precision therapy for PTCL.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with peripheral T-cell lymphoma (PTCL) by histopathology from June 2023 to December 2026 and detected by gene sequencing (NGS) with different molecular subtypes.
* Patients diagnosed with PTCL by histopathology from January 2023 to June 2023 and NGS detection can be performed if there is tumor tissue.
* Informed consented
* Age ≥ 18 years

Exclusion Criteria:

* History of malignancy except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix prior to study treatment
* Uncontrollable cardio-cerebral vascular, coagulative, autoimmune, serious infectious disease
* Not able to comply to the protocol for mental or other unknown reasons
* Patients with mentally disorders or other reasons unable to fully comply with the study protocol
* Pregnant or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators reviewed previous PTCL genomics and PTCL registry studies worldwide. And the number of PTCL patients admitted to each center per year was investigated. Sample of 1000 PTCL patients was suitable and able to obtain a statistical significant result.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-07-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Baseline up to data cut-off (up to approximately 2 years)
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
complete response rate | End of treatment visit (usually 6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Percentage of participants with complete response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Overall response rate | End of treatment visit (usually 6-8 weeks after last dose on Day 1 of Cycle 6 [Cycle length=21 days]
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria
Overall survival | Baseline up to data cut-off (up to approximately 4 years)
  Overall survival was defined as the time from the date of diagnosis to the date of death from any cause. Reported is the percentage of participants with event. of disease progression or relapse, using 2014 Lugano criteria,or death from any cause, whichever occurred first.
Duration of response | Baseline up to data cut-off (up to approximately 4 years)
  Time from first occurrence of documented CR or PR to disease progression/relapse, or death from any cause for participants with a response of CR or PR. Tumor assessments were performed with PET-CT.
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE | Baseline up to data cut-off (up to approximately 4 years)
  An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Tumor tissue gene mutations analysis | Baseline up to data cut-off (up to approximately 4 years)
  Targeted sequencing was used to detect 84 genes which can classify PTCL patients into different molecular subtypes.
Circulating free Deoxyribonucleic Acid (cfDNA) monitoring | Baseline up to data cut-off (up to approximately 4 years)
  CfDNA in peripheral blood assessed by local lab

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University People's Hospital, Beijing
  - Henan Cancer Hospital, Henan
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing
  - Department of Hematology, Shandong Provincial Hospital Affiliated to Shandong University, Jinan, China, Shandong
  - Shanghai Institute of Hematology, Rui-Jin Hospital affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Department of Hematology, West China Hospital, Sichuan University, Chengdu, Sichuan, China, Sichuan

IPD SHARING:
Plan to Share IPD: No